CLINICAL TRIAL: NCT02219932
Title: A Multicenter, Randomized, Double Blind, Placebo Controlled Study to Assess the Long-Term Efficacy and Safety of Prolonged Release Fampridine (BIIB041) 10 mg, Administered Twice Daily in Subjects With Multiple Sclerosis (ENHANCE)
Brief Title: Efficacy and Safety Study of Prolonged-Release Fampridine in Participants With Multiple Sclerosis
Acronym: ENHANCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 218MS305; 2013-003600-40 (EudraCT Number)
Record Dates: First submitted 2014-08-18; First posted 2014-08-19 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-01

CONDITIONS: Multiple Sclerosis
Keywords: Fampridine
MeSH Terms: conditions — Multiple Sclerosis | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fampridine 10 mg BID (Experimental): Prolonged-release fampridine 10 mg twice daily (BID) for up to 24 weeks
  Interventions: Drug: fampridine
- Placebo (Placebo Comparator): Matched placebo 10 mg BID for up to 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: fampridine
  Other Names: dalfampridine; Ampyra; Fampyra; fampridine prolonged-release tablets; BIIB041
  Arms: Fampridine 10 mg BID
Drug: Placebo — Matched placebo
  Arms: Placebo

SUMMARY:
The primary objective is to determine whether prolonged-release fampridine (10 mg twice daily) has a clinically meaningful effect on participant-reported walking ability over a 24-week study period.

The secondary objectives are: to determine whether prolonged-release fampridine 10 mg taken twice daily (BID) has a clinically meaningful effect on dynamic and static balance, physical impact of multiple sclerosis (MS), and upper extremity function over a 24-week study period; to evaluate criteria for early assessment of response to fampridine that can predict clinically meaningful benefits in walking ability and balance; to assess the safety and tolerability of prolonged-release fampridine 10 mg twice daily over a 24-week treatment period.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a diagnosis of primary-progressive, secondary-progressive, progressive-relapsing, or relapsing-remitting MS per revised McDonald Committee criteria [McDonald 2001; Polman 2005] as defined by Lublin and Reingold [Lublin and Reingold 1996] of at least 3 months duration
* Must have an Expanded Disability Status Scale (EDSS) score of 4 to 7, inclusive
* Must have walking impairment, as deemed by the Investigator

Key Exclusion Criteria:

* History of human immunodeficiency virus (HIV)
* Presence of acute or chronic hepatitis. Subjects who have evidence of prior hepatitis infection that has been serologically confirmed as resolved are not excluded from study participation
* Known allergy to fampridine, pyridine-containing substances, or any of the inactive ingredients in the prolonged-release fampridine tablet
* Creatinine clearance (CrCl) of <80 mL/min
* History of malignant disease
* Presence of pulmonary disease
* A body mass index (BMI) ≥40 (BMI formula: BMI = mass [kg]/[height(m)]2)

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 646 (Actual)
Dates: Start 2014-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (73):
- United States (15):
  - Research site, Cullman, Alabama
  - Research site, Phoenix, Arizona
  - Research site, San Diego, California
  - Research site, Bradenton, Florida
  - Research Site, Orlando, Florida
  - Research site, Tampa, Florida
  - Research site, West Palm Beach, Florida
  - Research site, Lexington, Kentucky
  - Research site, New Bedford, Massachusetts
  - Research site, Detroit, Michigan
  - Research site, Chesterfield, Missouri
  - Research site, Rochester, New York
  - Research site, Charlotte, North Carolina
  - Research site, Columbus, Ohio
  - Research site, Roanoke, Virginia
- Bulgaria (4):
  - Research site, Pleven
  - Research site, Plovdiv
  - Research site, Sofia
  - Research Site, Sofia
- Czechia (7):
  - Research site, Brno
  - Research site, Choceň
  - Research site, Havířov
  - Research site, Jihlava
  - Research site, Pardubice
  - Research site, Prague
  - Research site, Teplice
- Finland (4):
  - Research site, Helsinki
  - Research site, Oulu
  - Research site, Tampere
  - Research site, Turku
- Italy (5):
  - Research Site, Gallarate
  - Research site, Messina
  - Research site, Milan
  - Research site, Napoli
  - Research site, Rome
- Lithuania (3):
  - Research site, Kaunas
  - Research site, Klaipėda
  - Research site, Vilnius
- Netherlands (3):
  - Research Site, 's-Hertogenbosch
  - Research Site, Breda
  - Research Site, Sittard-Geleen
- Poland (12):
  - Research Site, Bialystok
  - Research site, Gdansk
  - Research site, Grudziądz
  - Research Site, Katowice
  - Research site, Katowice
  - Research Site, Kielce
  - Research site, Krakow
  - Research site, Lodz
  - Research site, Olsztyn
  - Research site, Plewiska
  - Research site, Rzeszów
  - Research site, Warsaw
- Russia (6):
  - Research Site, Kazan'
  - Research site, Kemerovo
  - Research site, Krasnoyarsk
  - Research Site, Moscow
  - Research site, Moscow
  - Research Site, Nizhny Novgorod
- Serbia (3):
  - Research site, Belgrade
  - Research site, Kragujevac
  - Research site, Niš
- United Kingdom (11):
  - Research site, Exeter, Devon
  - Research site, Plymouth, Devon
  - Research site, Romford, Essex
  - Research site, Salford, Greater Manchester
  - Research site, Norwich, Norfolk
  - Research site, Glasgow, Scotland
  - Research site, Chertsey, Surrey
  - Research site, Cardiff, Swansea
  - Research site, Birmingham, West Midlands
  - Research site, London
  - Research site, Nottingham

REFERENCES:
- [Derived] Hobart J, Ziemssen T, Feys P, Linnebank M, Goodman AD, Farrell R, Hupperts R, Blight AR, Englishby V, McNeill M, Chang I, Lima G, Elkins J; ENHANCE study investigators. Assessment of Clinically Meaningful Improvements in Self-Reported Walking Ability in Participants with Multiple Sclerosis: Results from the Randomized, Double-Blind, Phase III ENHANCE Trial of Prolonged-Release Fampridine. CNS Drugs. 2019 Jan;33(1):61-79. doi: 10.1007/s40263-018-0586-5. PMID 30535670

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 646 participants were enrolled. A single site in Poland was later closed due to serious Good Clinical Practice noncompliance issues observed during the conduct of the study. There were 10 participants randomized at this site (6 to fampridine and 4 to placebo). The data from this site were excluded from all analyses.
Groups:
- Placebo: Placebo twice daily (BID) for up to 24 weeks
- Fampridine 10 mg BID: Prolonged-release fampridine 10 mg BID for up to 24 weeks
Period: Overall Study
Arm/Group | Placebo | Fampridine 10 mg BID
Started | 319 | 317
Randomized, Not Treated | 0 | 1
Completed | 254 | 266
Not Completed | 65 | 51
Not completed — Other | 5 | 11
Not completed — Death | 1 | 1
Not completed — Investigator Decision | 0 | 1
Not completed — Consent Withdrawn | 11 | 7
Not completed — Lack of Efficacy (Subject Perception) | 10 | 2
Not completed — Protocol Violation | 10 | 6
Not completed — Pregnancy | 1 | 0
Not completed — Lost to Follow-up | 4 | 2
Not completed — Adverse Event | 23 | 21

BASELINE CHARACTERISTICS:
Population: Safety population: all participants who received at least 1 dose of study drug.
Groups:
- Placebo: Placebo BID for up to 24 weeks
- Total: Total of all reporting groups
Arm/Group | Placebo | Fampridine 10 mg BID | Total
Number analyzed (Participants) | 319 | 316 | 635
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (10.50) | 49.0 (9.82) | 48.9 (10.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 181 | 187 | 368
  Male | 138 | 129 | 267

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Achieving a Mean Improvement of ≥ 8 Points From Baseline on the Multiple Sclerosis Walking Scale (MSWS-12) Over 24 Weeks
Description: MSWS-12 is a participant self-assessment of the walking limitations due to MS during the past 2 weeks. It contains 12 items that measure the impact of MS on walking. Items are summed to generate a total score and transformed to a scale with a range of 0 to 100, where higher scores indicate greater impact on walking.
  A responder is defined as a participant with a mean improvement of at least 8 points over 24 weeks compared to baseline. Baseline is defined as the mean at Screening and Day 1 visits. If a participant has a mean MSWS-12 score of < 0.5 over the double-blind period, and a baseline MSWS-12 score of < 8 points, the participant is counted as a responder. A participant who indicates they cannot walk at all on MSWS-12 during any double-blind visit, and who shows severe disability and an inability to walk on other efficacy assessments is counted as a non-responder. Estimated proportion obtained from binomial proportions.
Time Frame: Baseline to 24 weeks
Population: Intent-to-treat population: participants who received at least 1 dose of study drug and had at least 1 postbaseline efficacy assessment.
Measure: Number; unit: proportion of participants
Arm/Group | Placebo | Fampridine 10 mg BID
Number analyzed (Participants) | 318 | 315
proportion of participants | 0.336 | 0.432
Statistical Analysis 1: Comparison: Placebo vs Fampridine 10 mg BID; Based on logistic regression, adjusting for baseline MSWS-12 score, baseline TUG speed, age, screening Expanded Disability Status Scale (EDSS) score and prior aminopyridine. Missing data handled by multiple imputation. Hypothesis testing was performed at the 2-sided 5% significance level overall, with adjustment for testing multiple secondary endpoints; Test type: Superiority or Other; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 1.61, 95% CI 2-sided [1.15 to 2.26] — fampridine vs. placebo
Statistical Analysis 2: Comparison: Placebo vs Fampridine 10 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Risk Difference for Adjusted Proportions = 0.104, 95% CI 2-sided [0.030 to 0.178]
Statistical Analysis 3: Comparison: Placebo vs Fampridine 10 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Relative Risk = 1.38, 95% CI 2-sided [1.06 to 1.70]

2. Secondary Outcome: Proportion of Participants Achieving a Mean Improvement From Baseline of ≥ 15% in Timed Up and Go (TUG) Speed Over 24 Weeks
Description: TUG is a timed walking test designed to measure gait performance and balance. It measures in seconds the time taken by an individual to stand up from a standard arm chair (approximate seat height of 46 cm [18in], arm height 65 cm [25.6 in]), walk a distance of 3 meters (118 inches, approximately 10 feet), turn, walk back to the chair, and sit down.
  A responder is defined as a participant with a mean improvement of at least 15% in TUG speed over 24 weeks compared to baseline. Baseline is defined as the mean at Screening and Day 1 visits. Estimated proportion obtained from binomial proportions. There are 2 TUG tests given, and the average across the 2 tests is used to calculate average speed. Healthy participants below the age of 79 are expected to complete this task in 7-10 seconds (American College of Rheumatology). Missing data are handled using multiple imputation and baseline is defined as the mean over Screening and Day 1.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Number; unit: proportion of participants
Arm/Group | Placebo | Fampridine 10 mg BID
Number analyzed (Participants) | 318 | 315
proportion of participants | 0.347 | 0.434
Statistical Analysis 1: Comparison: Placebo vs Fampridine 10 mg BID; Based on logistic regression, adjusting for baseline TUG speed, screening EDSS score and prior aminopyridine. Missing data were handled using multiple imputation; Test type: Superiority or Other; p = 0.030, Regression, Logistic; Odds Ratio (OR) = 1.46, 95% CI 2-sided [1.04 to 2.07]
Statistical Analysis 2: Comparison: Placebo vs Fampridine 10 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Risk Difference for Adjusted Proportions = 0.092, 95% CI 2-sided [0.009 to 0.175]
Statistical Analysis 3: Comparison: Placebo vs Fampridine 10 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Relative Risk = 1.25, 95% CI 2-sided [0.99 to 1.51]

3. Secondary Outcome: Change From Baseline in Multiple Sclerosis Impact Scale-29 (MSIS-29) Physical Score Over 24 Weeks
Description: The 29-item MSIS-29 is a participant-reported outcome measure to assess the impact of MS on day-to-day life during the past 2 weeks from a participant's perspective; it measures 20 physical items and 9 psychological items. The physical score is generated by summing individual items and then transforming to a scale with a range of 0 (no impact of MS) to 100 (extreme impact of MS); a negative change indicates an improvement in function.
  Data are based on a mixed model for repeated measures (MMRM) model using a common variance AR(1) variance-covariance matrix structure. Treatment, visit and treatment by visit interaction were included in the model as explanatory variables, adjusting for screening EDSS, baseline MSIS-29 physical score and prior aminopyridine as covariates. Missing data are handled using multiple imputation and baseline is defined as the mean over screening and Day 1.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Fampridine 10 mg BID
Number analyzed (Participants) | 318 | 315
units on a scale | -4.68 (0.936) | -8.00 (0.911)
Statistical Analysis 1: Comparison: Placebo vs Fampridine 10 mg BID; Test type: Superiority or Other; p < 0.001, mixed model for repeated measures; LS Mean Difference = -3.31, 95% CI 2-sided [-5.13 to -1.50], Standard Error of Mean 0.925

4. Secondary Outcome: Change From Baseline in Berg Balance Scale (BBS) Over 24 Weeks
Description: The BBS is a widely used assessment tool to identify balance impairment. Functional activities such as reaching, bending, transferring, and standing are evaluated on the test to evaluate balance. Participants are asked to complete 14 tasks that are rated from 0 (cannot perform) to 4 (normal performance) for a total of 56 points. BBS scores range from 0 (poor balance) to 56 (good balance); a positive change indicates improvement.
  Data are based on an MMRM model using a common variance AR(1) variance-covariance matrix structure. Treatment, visit and treatment by visit interaction were included in the model as explanatory variables, adjusting for screening EDSS, baseline BBS and prior aminopyridine as covariates. Missing data are handled using multiple imputation and baseline is defined as the mean over screening and Day 1.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Fampridine 10 mg BID
Number analyzed (Participants) | 318 | 315
units on a scale | 1.34 (0.284) | 1.75 (0.278)
Statistical Analysis 1: Comparison: Placebo vs Fampridine 10 mg BID; Test type: Superiority or Other; p = 0.141, mixed model for repeated measures; LS Mean Difference = 0.41, 95% CI 2-sided [-0.13 to 0.95], Standard Error of Mean 0.277

5. Secondary Outcome: Change From Baseline in ABILHAND Score Over 24 Weeks
Description: The ABILHAND Questionnaire measures a participant's perceived difficulty in performing everyday manual activities in the last 3 months. The participant completes a 56-item questionnaire by estimating their own difficulty or ease in performing each of 56 activities. Items are summed to generate a total score and transformed to a scale with a range of 0 (poor manual ability) to 100 (good manual ability); a positive change indicates an improvement in manual ability.
  Data are based on an MMRM model using a common variance AR(1) variance-covariance matrix structure. Treatment, visit and treatment by visit interaction were included in the model as explanatory variables, adjusting for screening EDSS, baseline ABILHAND and prior aminopyridine as covariates. Missing data are handled using multiple imputation and baseline is defined as the Day 1 assessment.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population: participants who received at least 1 dose of study drug and had at least 1 postbaseline efficacy assessment and available data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Fampridine 10 mg BID
Number analyzed (Participants) | 315 | 312
units on a scale | 0.75 (0.593) | 1.49 (0.574)
Statistical Analysis 1: Comparison: Placebo vs Fampridine 10 mg BID; Test type: Superiority or Other; p = 0.197, mixed model for repeated measures; LS Mean Difference = 0.74, 95% CI 2-sided [-0.38 to 1.86], Standard Error of Mean 0.573

ADVERSE EVENTS:
Time Frame: Collected through follow-up (14 [±3] days following Week 24/Early Termination). Serious adverse events collected from signing of informed consent; adverse events collected from first dose of study treatment.
Groups:
- Fampridine 10mg BID: Prolonged-release fampridine 10 mg BID for up to 24 weeks
Arm/Group | Placebo | Fampridine 10mg BID
Serious Adverse Events (participants affected / at risk) | 21/319 | 25/316
Other Adverse Events (participants affected / at risk) | 93/319 | 100/316
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=319) | Fampridine 10mg BID (N=316)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Gallbladder empyema (Infections and infestations) | 0 | 1
Injection site infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 2
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian endometrioid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Multiple sclerosis relapse (Nervous system disorders) | 10 | 14
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0
Endometrial atrophy (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=319) | Fampridine 10mg BID (N=316)
Nasopharyngitis (Infections and infestations) | 18 | 15
Urinary tract infection (Infections and infestations) | 29 | 40
Fall (Injury, poisoning and procedural complications) | 17 | 22
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 16
Multiple sclerosis relapse (Nervous system disorders) | 31 | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.